CLINICAL TRIAL: NCT02735200
Title: Topical Delivery of Vitamin D3: A Randomized Controlled Trial (RCT)
Brief Title: Topical Delivery of Vitamin D3 as Vitamin D Supplementation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DammamU
Record Dates: First submitted 2016-03-12; First posted 2016-04-12 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: assignment
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topical Vitamin D3 application (Experimental): Intervention is Application of topical Vitamin D3 Frequency: Daily Dosage: 1 gram (5000 IU) Duration: 120 days
  Interventions: Drug: Application of topical vitamin d3 (Top-D)
- Aloe vera gel Application (Active Comparator): Application of Aloe vera gel will be carried out Dosage: 1 gram Frequency: Daily Duration: 120 days
  Interventions: Other: Application of Aloe vera gel

INTERVENTIONS:
Drug: Application of topical vitamin d3 (Top-D) — Topical Vitamin D3 will be applied on the skin, externally, 1 gram daily for 120 days
  Other Names: Topical vitamin D3; TOP-D
  Arms: Topical Vitamin D3 application
Other: Application of Aloe vera gel — aloe vera gel will be applied
  Dosage: 1 gram Duration: 120 days Frequency: Daily
  Arms: Aloe vera gel Application

SUMMARY:
After obtaining the approval from the IRB of University of Dammam and informed consent from 550 healthy patients, with vitamin D deficiency and vitamin D insufficiency and deficiency were recruited. Age, weight and height will be taken, a detailed history, meticulous clinical examination was performed to rule out any diseases and complete blood picture, serum calcium, phosphorous, alkaline phosphatase, Parathormone and 25 Hydroxy-vitamin D (25OHD) will be done. 25-Hydroxy Vitamin D3 was measured in house by chemiluminescence immunoassay (CLIA) and ≥30ng/mL was taken as normal, 21-29ng/mL as insufficiency and ≤20 ng/mL as deficiency. The participants were divided into two groups of 350 in study arm and 200 in control arm. All participants were instructed not to change their dietary habits and life style till the study was over. The study group of women were instructed to apply to apply Top-D (Proniosomal Delivered- Vitamin D3) 1 gram containing 5000 IU of vitamin D3. The second group used 1 gram of Aloe vera gel. The participants had no knowledge to which group they belong. A second blood sample was taken at the end of 4 months and the data was entered in the data base and analyzed using SPSS Inc version 19.

DETAILED DESCRIPTION:
After obtaining the approval from the Institutional Review Board (IRB) of University of Dammam and informed consent from 550 healthy patients, with vitamin D deficiency and vitamin D insufficiency and deficiency were recruited. Age, weight and height will be taken, a detailed history, meticulous clinical examination was performed to rule out any diseases and complete blood picture, serum calcium, phosphorous, alkaline phosphatase, Parathormone and 25 Hydroxy-vitamin D (25OHD) will be done. 25-Hydroxy Vitamin D3 was measured in house by chemiluminescence immunoassay (CLIA) and ≥30ng/mL was taken as normal, 21-29ng/mL as insufficiency and ≤20 ng/mL as deficiency. The participants were divided into two groups of 350 in study arm and 200 in control arm. All participants were instructed not to change their dietary habits and life style till the study was over. The study group of women were instructed to apply to apply Top-D (Proniosomal Delivered- Vitamin D3) I gram gram containing 5000 IU of vitamin D3. The second group used 1 gram of Aloe vera gel. The participants had no knowledge to which group they belong. A second blood sample was taken at the end of 4 months and the data was entered in the data base and analyzed using SPSS Inc version 19.

ELIGIBILITY:
Inclusion Criteria:

all men and women with vitamin D insufficiency and deficiency Must be able to apple the topical vitamin D3 Must be willing to sign and informed consent

Exclusion Criteria:

* Those who have normal 25OHD levels

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2016-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naif AlMasoud, MD, PhD, Study Director — University of Dammam, Saudi Arabia
Locations (1):
- King Fahd Hospital of the University, Khobar, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Riccio PA, Zingaretti C, Milani M, Ricci Petitoni G, Monti G, Pavanello PM. [Thymoma: diagnosis and surgical treatment]. Minerva Chir. 1996 Sep;51(9):663-7. Italian. PMID 9082230
- [Background] Sadat-Ali M, AlElq A, Al-Turki H, Al-Mulhim F, Al-Ali A. Vitamin D levels in healthy men in eastern Saudi Arabia. Ann Saudi Med. 2009 Sep-Oct;29(5):378-82. doi: 10.4103/0256-4947.55168. PMID 19700896
- [Background] Elsammak MY, Al-Wosaibi AA, Al-Howeish A, Alsaeed J. Vitamin d deficiency in Saudi Arabs. Horm Metab Res. 2010 May;42(5):364-8. doi: 10.1055/s-0030-1248296. Epub 2010 Mar 8. PMID 20213587
- [Background] Al-Elq AH. The status of Vitamin D in medical students in the preclerkship years of a Saudi medical school. J Family Community Med. 2012 May;19(2):100-4. doi: 10.4103/2230-8229.98293. PMID 22870413
- [Background] Grant AM, Avenell A, Campbell MK, McDonald AM, MacLennan GS, McPherson GC, Anderson FH, Cooper C, Francis RM, Donaldson C, Gillespie WJ, Robinson CM, Torgerson DJ, Wallace WA; RECORD Trial Group. Oral vitamin D3 and calcium for secondary prevention of low-trauma fractures in elderly people (Randomised Evaluation of Calcium Or vitamin D, RECORD): a randomised placebo-controlled trial. Lancet. 2005 May 7-13;365(9471):1621-8. doi: 10.1016/S0140-6736(05)63013-9. PMID 15885294
- [Background] Porthouse J, Cockayne S, King C, Saxon L, Steele E, Aspray T, Baverstock M, Birks Y, Dumville J, Francis R, Iglesias C, Puffer S, Sutcliffe A, Watt I, Torgerson DJ. Randomised controlled trial of calcium and supplementation with cholecalciferol (vitamin D3) for prevention of fractures in primary care. BMJ. 2005 Apr 30;330(7498):1003. doi: 10.1136/bmj.330.7498.1003. PMID 15860827
- [Background] Jackson RD, LaCroix AZ, Gass M, Wallace RB, Robbins J, Lewis CE, Bassford T, Beresford SA, Black HR, Blanchette P, Bonds DE, Brunner RL, Brzyski RG, Caan B, Cauley JA, Chlebowski RT, Cummings SR, Granek I, Hays J, Heiss G, Hendrix SL, Howard BV, Hsia J, Hubbell FA, Johnson KC, Judd H, Kotchen JM, Kuller LH, Langer RD, Lasser NL, Limacher MC, Ludlam S, Manson JE, Margolis KL, McGowan J, Ockene JK, O'Sullivan MJ, Phillips L, Prentice RL, Sarto GE, Stefanick ML, Van Horn L, Wactawski-Wende J, Whitlock E, Anderson GL, Assaf AR, Barad D; Women's Health Initiative Investigators. Calcium plus vitamin D supplementation and the risk of fractures. N Engl J Med. 2006 Feb 16;354(7):669-83. doi: 10.1056/NEJMoa055218. PMID 16481635
- [Background] Nikolaus T, Kruse W, Bach M, Specht-Leible N, Oster P, Schlierf G. Elderly patients' problems with medication. An in-hospital and follow-up study. Eur J Clin Pharmacol. 1996;49(4):255-9. doi: 10.1007/BF00226324. PMID 8857069
- [Background] Thomas BJ, Finnin BC. The transdermal revolution. Drug Discov Today. 2004 Aug 15;9(16):697-703. doi: 10.1016/S1359-6446(04)03180-0. PMID 15341783
- [Background] Shi Y, Wei Z, Zhao H, Liu T, Dong A, Zhang J. Electrospinning of ibuprofen-loaded composite nanofibers for improving the performances of transdermal patches. J Nanosci Nanotechnol. 2013 Jun;13(6):3855-63. doi: 10.1166/jnn.2013.7157. PMID 23862418
- [Background] Derry S, Moore RA. Topical capsaicin (low concentration) for chronic neuropathic pain in adults. Cochrane Database Syst Rev. 2012 Sep 12;2012(9):CD010111. doi: 10.1002/14651858.CD010111. PMID 22972149
- [Background] Aggarwal N, Goindi S. Preparation and in vivo evaluation of solid lipid nanoparticles of griseofulvin for dermal use. J Biomed Nanotechnol. 2013 Apr;9(4):564-76. doi: 10.1166/jbn.2013.1569. PMID 23621015
- [Background] Ahad A, Al-Jenoobi FI, Al-Mohizea AM, Aqil M, Kohli K. Transdermal delivery of calcium channel blockers for hypertension. Expert Opin Drug Deliv. 2013 Aug;10(8):1137-53. doi: 10.1517/17425247.2013.783562. Epub 2013 Mar 26. PMID 23527660
- [Background] Goodman MP. Are all estrogens created equal? A review of oral vs. transdermal therapy. J Womens Health (Larchmt). 2012 Feb;21(2):161-9. doi: 10.1089/jwh.2011.2839. Epub 2011 Oct 19. PMID 22011208
- [Background] Segal E, Zinman C, Raz B, Ish-Shalom S. Low patient compliance--a major negative factor in achieving vitamin D adequacy in elderly hip fracture patients supplemented with 800IU of vitamin D3 daily. Arch Gerontol Geriatr. 2009 Nov-Dec;49(3):364-7. doi: 10.1016/j.archger.2008.12.001. Epub 2009 Jan 14. PMID 19147237
- [Background] Castelo-Branco C, Cortes X, Ferrer M; UNICAD study investigators. Treatment persistence and compliance with a combination of calcium and vitamin D. Climacteric. 2010 Dec;13(6):578-84. doi: 10.3109/13697130903452804. Epub 2009 Dec 1. PMID 19951084
- [Background] Sanfelix-Genoves J, Gil-Guillen VF, Orozco-Beltran D, Giner-Ruiz V, Pertusa-Martinez S, Reig-Moya B, Carratala C. Determinant factors of osteoporosis patients' reported therapeutic adherence to calcium and/or vitamin D supplements: a cross-sectional, observational study of postmenopausal women. Drugs Aging. 2009;26(10):861-9. doi: 10.2165/11317070-000000000-00000. PMID 19761279
- [Result] Sadat-Ali M, Bubshait DA, Al-Turki HA, Al-Dakheel DA, Al-Olayani WS. Topical delivery of vitamin d3: a randomized controlled pilot study. Int J Biomed Sci. 2014 Mar;10(1):21-4. PMID 24711745

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Orthopedic clinics
Pre-assignment Details: consecutive patients
Groups:
- Application of Aloe Vera Gel: Intervention: aloe vera gel administration was applied 1 gram daily for 120 days.
- Topical Application of Vitamin D3: topical vitamin D3 in intervention group: local application of Top-D, 1 gram (5000 IU) was applied every day, for 120 days.
Period: Overall Study
Arm/Group | Application of Aloe Vera Gel | Topical Application of Vitamin D3
Started | 200 | 350
Completed | 192 | 345
Not Completed | 8 | 5
Not completed — Lost to Follow-up | 0 | 5
Not completed — Withdrawal by Subject | 8 | 0

BASELINE CHARACTERISTICS:
Groups:
- Topical Application of Vitamin D3: this arm received topical vitamin D3 1gram (5000IU)
- Application of Aloe Vera Gel: Intervention: aloe vera gel administration 1 gram
- Total: Total of all reporting groups
Arm/Group | Topical Application of Vitamin D3 | Application of Aloe Vera Gel | Total
Number analyzed (Participants) | 350 | 200 | 550
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 300 | 171 | 471
  >=65 years | 50 | 29 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.59 (15.74) | 41.6 (16.6) | 41.9 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 285 | 137 | 422
  Male | 65 | 63 | 128
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Saudi Arabia | 350 | 200 | 550

OUTCOME MEASURES:

1. Primary Outcome: Level of Serum 25 OHD Level Pre-treatment and Post Treatment
Description: Patients had analysis of serum 25 OHD level pre and post treatment, to check if treatment with Topical Vitamin D made any difference.
Time Frame: baseline and 5 months
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Topical Application of Vitamin D3: Intervention: patients will be administered topical vitamin D3 5000 IU
  topical vitamin D3 in intervention group: local application
- Application of Aloe Vera Gel: Intervention: aloe vera gel administration
Arm/Group | Topical Application of Vitamin D3 | Application of Aloe Vera Gel
Number analyzed (Participants) | 345 | 192
ng/mL
  pre treatment | 12.03 (4.57) | 10.36 (4.09)
  post treatment | 37.17 (6.04) | 10.51 (3.5)
Statistical Analysis 1: Comparison: Topical Application of Vitamin D3 vs Application of Aloe Vera Gel; Test type: Superiority; p = 0.9, t-test, 2 sided — the p value correspond to the pretreatment time frame; Mean Difference (Final Values) = 1.67
Statistical Analysis 2: Comparison: Topical Application of Vitamin D3 vs Application of Aloe Vera Gel; Test type: Superiority; p < 0.001, t-test, 2 sided — p value corresponds to the post treatment time frame; Mean Difference (Final Values) = 26.66

ADVERSE EVENTS:
Groups:
- Application of Aloe Vera Gel: Intervention: aloe vera gel administration
  topical vitamin D3 in intervention group: local application
Arm/Group | Topical Application of Vitamin D3 | Application of Aloe Vera Gel
All-Cause Mortality (participants affected / at risk) | 0/345 | 0/192
Serious Adverse Events (participants affected / at risk) | 0/345 | 0/192
Other Adverse Events (participants affected / at risk) | 0/345 | 0/192

LIMITATIONS AND CAVEATS:
we did have a limitation of not performing the absorption studies, which could have strenthened the study robustly.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes